CLINICAL TRIAL: NCT02628067
Title: A Clinical Trial of Pembrolizumab (MK-3475) Evaluating Predictive Biomarkers in Subjects With Advanced Solid Tumors (KEYNOTE 158)
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Advanced Solid Tumors (MK-3475-158/KEYNOTE-158)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-158; 163196 (Registry Identifier: JAPIC-CTI); MK-3475-158 (Other: MSD); KEYNOTE-158 (Other: MSD); 2022-501253-37-00 (Registry Identifier: EU CT); U1111-1275-8374 (Registry Identifier: UTN); 2015-002067-41 (EudraCT Number)
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancer; Anal Carcinoma; Anal Cancer; Biliary Cancer; Cholangiocarcinoma; Bile Duct Cancer; Neuroendocrine Tumor; Carcinoid Tumor; Endometrial Carcinoma; Endometrial Cancer; Cervical Carcinoma; Cervical Cancer; Vulvar Carcinoma; Vulvar Cancer; Small Cell Lung Carcinoma; Small Cell Lung Cancer (SCLC); Mesothelioma; Thyroid Carcinoma; Thyroid Cancer; Salivary Gland Carcinoma; Salivary Gland Cancer; Salivary Cancer; Parotid Gland Cancer; Advanced Solid Tumors; Colorectal Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); microsatellite instability (MSI); mismatch repair (MMR)
MeSH Terms: conditions — Anus Neoplasms; Biliary Tract Neoplasms; Cholangiocarcinoma; Bile Duct Neoplasms; Neuroendocrine Tumors; Carcinoid Tumor; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Small Cell Lung Carcinoma; Mesothelioma; Thyroid Neoplasms; Salivary Gland Neoplasms; Parotid Neoplasms; Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body; Microsatellite Instability | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab 200 mg (Experimental): Participants will receive pembrolizumab 200 mg intravenously on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years of treatment).
  Interventions: Biological: pembrolizumab
- Pembrolizumab 400 mg (Experimental): Participants with any advanced solid tumor that has failed at least one line of therapy and is Tumor- Mutational Burden-High (TMB-H), excluding participants with mismatch repair deficient (dMMR/MSI-H) tumors. The dosing regimen for this cohort will be 400 mg every 6 weeks (Q6W) for up to 18 administrations (up to approximately 2 years of treatment).
  Interventions: Biological: pembrolizumab

INTERVENTIONS:
Biological: pembrolizumab — intravenous infusion
  Other Names: MK-3475; SCH 900475; KEYTRUDA®
  Arms: Pembrolizumab 200 mg
Biological: pembrolizumab — intravenous infusion
  Other Names: MK-3475; SCH 900475; KEYTRUDA®
  Arms: Pembrolizumab 400 mg

SUMMARY:
In this study, participants with multiple types of advanced (unresectable and/or metastatic) solid tumors who have progressed on standard of care therapy will be treated with pembrolizumab (MK-3475).

ELIGIBILITY:
Inclusion Criteria:

- Histologically or cytologically-documented, advanced solid tumor of one of the following types:

* Anal Squamous Cell Carcinoma
* Biliary Adenocarcinoma (gallbladder or biliary tree (intrahepatic or extrahepatic cholangiocarcinoma) except Ampulla of Vater cancers)
* Neuroendocrine Tumors (well- and moderately-differentiated) of the lung, appendix, small intestine, colon, rectum, or pancreas
* Endometrial Carcinoma (sarcomas and mesenchymal tumors are excluded)
* Cervical Squamous Cell Carcinoma
* Vulvar Squamous Cell Carcinoma
* Small Cell Lung Carcinoma
* Mesothelioma
* Thyroid Carcinoma
* Salivary Gland Carcinoma (sarcomas and mesenchymal tumors are excluded)
* Any advanced solid tumor, with the exception of colorectal carcinoma (CRC), which is Microsatellite Instability (MSI)-High (MSI-H) OR
* Any advanced solid tumor (including Colorectal Carcinoma [CRC]) which is Mismatch Repair Deficient (dMMR)/MSI-H in participants from mainland China who are of Chinese descent. (CRC participants will have a histologically proven locally advanced unresectable or metastatic CRC which is dMMR/MSI-H that has received 2 prior lines of therapy) OR
* Any advanced solid tumor that has failed at least one line of therapy and is TMB-H (≥10 mut/Mb, F1CDx assay), excluding dMMR/MSI-H tumors.

Note: For participants to be eligible for enrollment they must have failed at least one line of standard of care systemic therapy (ie, not treatment naïve), with the exception of CRC participants who must have failed at least 2 lines of standard of care systemic therapy, as per CRC specific eligibility criteria. Participants must not have melanoma or NSCLC.

* Progression of tumor or intolerance to therapies known to provide clinical benefit. There is no limit to the number of prior treatment regimens
* Can supply tumor tissue for study analyses (dependent on tumor type)
* Radiologically-measurable disease
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale within 3 days prior to first dose of pembrolizumab
* Life expectancy of at least 3 months
* Adequate organ function
* Female participants of childbearing potential must be willing to use adequate contraception during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention. and agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period. The length of time required to continue contraception for each study intervention is as follows: MK-3475 (120 days)

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study treatment
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or not recovered from an adverse event caused by mAbs administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks of study Day 1 or not recovered from adverse events caused by a previously administered agent
* Known additional malignancy within 2 years prior to enrollment with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cancers
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has known glioblastoma multiforme of the brain stem
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with the participant's ability to cooperate with the requirements of the study
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Previously participated in any other pembrolizumab (MK-3475) study, or received prior therapy with an anti-programmed cell death (PD)-1, anti-PD-Ligand 1 (anti-PD-L1), anti-PD-Ligand 2 (anti-PD-L2), or any other immunomodulating mAb or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Known history of Human Immunodeficiency Virus (HIV)
* Known active Hepatitis B or C
* Received live vaccine within 30 days of planned start of study treatment
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Known history of active tuberculosis (TB, Bacillus tuberculosis)
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1609 (Estimated)
Dates: Start 2015-12-18 (Actual); Primary Completion 2027-05-04 (Estimated); Study Completion 2027-05-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 10.5 years
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ at any time during the trial. Responses will be determined by independent central radiologic review, with confirmatory assessment as required per RECIST 1.1. Participants with unknown or missing response information will be treated as non-responders. The percentage of participants who experience a CR or PR based on modified RECIST 1.1 will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 10.5 years
  DOR, defined in the subset of participants with a CR or PR, based on RECIST 1.1 as assessed by independent central radiologic review, as the time from first documented evidence of CR or PR until the first documented sign of disease progression or death due to any cause, whichever occurs first. A Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. Participants who are alive, have not progressed, have not initiated new anti-cancer treatment, and have not been determined to be lost to follow-up are considered ongoing responders at the time of analysis.
Progression Free Survival (PFS) | Up to approximately 10.5 years
  PFS is defined as the time from allocation to the first documented disease progression according to RECIST 1.1 as assessed by independent central radiologic review, or death due to any cause, whichever occurs first. Per RECIST 1.1, progressive disease (PD) is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. If a participant does not have a documented date of progression or death, PFS will be censored at the date of the last adequate assessment.
Overall Survival (OS) | Up to approximately 10.5 years
  OS is defined as the time from randomization to death due to any cause. OS will be presented. Censoring will be performed using the date of last known contact for those who are alive at the time of analysis.
Percentage of Participants with Adverse Events (AEs) | Up to approximately 27 months
  An adverse event (AE) is defined as any untoward medical occurrence in a study participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this intervention. The percentage of participants with AEs will be reported.
Percentage of Participants who Discontinue Study Intervention due to AEs | Up to approximately 2 years
  An AE is defined as any untoward medical occurrence in a study participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. The percentage of participants who discontinue study intervention due to AEs will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Marabelle A, Le DT, Ascierto PA, Di Giacomo AM, De Jesus-Acosta A, Delord JP, Geva R, Gottfried M, Penel N, Hansen AR, Piha-Paul SA, Doi T, Gao B, Chung HC, Lopez-Martin J, Bang YJ, Frommer RS, Shah M, Ghori R, Joe AK, Pruitt SK, Diaz LA Jr. Efficacy of Pembrolizumab in Patients With Noncolorectal High Microsatellite Instability/Mismatch Repair-Deficient Cancer: Results From the Phase II KEYNOTE-158 Study. J Clin Oncol. 2020 Jan 1;38(1):1-10. doi: 10.1200/JCO.19.02105. Epub 2019 Nov 4. PMID 31682550
- [Result] Marabelle A, O'Malley DM, Hendifar AE, Ascierto PA, Motola-Kuba D, Penel N, Cassier PA, Bariani G, De Jesus-Acosta A, Doi T, Longo F, Miller WH Jr, Oh DY, Gottfried M, Yao L, Jin F, Gozman A, Maio M. Pembrolizumab in microsatellite-instability-high and mismatch-repair-deficient advanced solid tumors: updated results of the KEYNOTE-158 trial. Nat Cancer. 2025 Feb;6(2):253-258. doi: 10.1038/s43018-024-00894-y. Epub 2025 Feb 20. PMID 39979665
- [Derived] Wu X, Mao Y, Xu N, Bai Y, Wang D, Chen X, Yin X, Deng Y, Yang J, Zhang J, Tang J, Huang Y, Li J, Luo S, Zheng H, Zhao W, Xu M, Li N, Mao Y, Gozman A, Xu J. Pembrolizumab in Patients of Chinese Descent with Microsatellite Instability-high/Mismatch Repair Deficient Advanced Solid Tumors: KEYNOTE-158 Final Analysis. Adv Ther. 2025 May;42(5):2480-2489. doi: 10.1007/s12325-025-03142-6. Epub 2025 Mar 22. PMID 40121391
- [Derived] Oh DY, Algazi A, Capdevila J, Longo F, Miller W Jr, Chun Bing JT, Bonilla CE, Chung HC, Guren TK, Lin CC, Motola-Kuba D, Shah M, Hadoux J, Yao L, Jin F, Norwood K, Lebellec L. Efficacy and safety of pembrolizumab monotherapy in patients with advanced thyroid cancer in the phase 2 KEYNOTE-158 study. Cancer. 2023 Apr 15;129(8):1195-1204. doi: 10.1002/cncr.34657. Epub 2023 Feb 7. PMID 36748723
- [Derived] O'Malley DM, Bariani GM, Cassier PA, Marabelle A, Hansen AR, De Jesus Acosta A, Miller WH Jr, Safra T, Italiano A, Mileshkin L, Amonkar M, Yao L, Jin F, Norwood K, Maio M. Health-related quality of life with pembrolizumab monotherapy in patients with previously treated advanced microsatellite instability high/mismatch repair deficient endometrial cancer in the KEYNOTE-158 study. Gynecol Oncol. 2022 Aug;166(2):245-253. doi: 10.1016/j.ygyno.2022.06.005. Epub 2022 Jul 11. PMID 35835611
- [Derived] Even C, Delord JP, Price KA, Nakagawa K, Oh DY, Burge M, Chung HC, Doi T, Fakih M, Takahashi S, Yao L, Jin F, Norwood K, Hansen AR. Evaluation of pembrolizumab monotherapy in patients with previously treated advanced salivary gland carcinoma in the phase 2 KEYNOTE-158 study. Eur J Cancer. 2022 Aug;171:259-268. doi: 10.1016/j.ejca.2022.05.007. Epub 2022 Jun 28. PMID 35777186
- [Derived] Maio M, Ascierto PA, Manzyuk L, Motola-Kuba D, Penel N, Cassier PA, Bariani GM, De Jesus Acosta A, Doi T, Longo F, Miller WH, Oh DY, Gottfried M, Xu L, Jin F, Norwood K, Marabelle A. Pembrolizumab in microsatellite instability high or mismatch repair deficient cancers: updated analysis from the phase II KEYNOTE-158 study. Ann Oncol. 2022 Sep;33(9):929-938. doi: 10.1016/j.annonc.2022.05.519. Epub 2022 Jun 6. PMID 35680043
- [Derived] Maio M, Amonkar MM, Norquist JM, Ascierto PA, Manzyuk L, Motola-Kuba D, Penel N, Cassier PA, Bariani GM, De Jesus Acosta A, Doi T, Longo F, Miller WH Jr, Oh DY, Gottfried M, Wang R, Norwood K, Marabelle A. Health-related quality of life in patients treated with pembrolizumab for microsatellite instability-high/mismatch repair-deficient advanced solid tumours: Results from the KEYNOTE-158 study. Eur J Cancer. 2022 Jul;169:188-197. doi: 10.1016/j.ejca.2022.03.040. Epub 2022 May 16. PMID 35588692
- [Derived] Shapira-Frommer R, Mileshkin L, Manzyuk L, Penel N, Burge M, Piha-Paul SA, Girda E, Lopez Martin JA, van Dongen MGJ, Italiano A, Xu L, Jin F, Norwood K, Ott PA. Efficacy and safety of pembrolizumab for patients with previously treated advanced vulvar squamous cell carcinoma: Results from the phase 2 KEYNOTE-158 study. Gynecol Oncol. 2022 Aug;166(2):211-218. doi: 10.1016/j.ygyno.2022.01.029. Epub 2022 Mar 28. PMID 35361487
- [Derived] Marabelle A, Cassier PA, Fakih M, Kao S, Nielsen D, Italiano A, Guren TK, van Dongen MGJ, Spencer K, Bariani GM, Ascierto PA, Santoro A, Shah M, Asselah J, Iqbal S, Takahashi S, Piha-Paul SA, Ott PA, Chatterjee A, Jin F, Norwood K, Delord JP. Pembrolizumab for previously treated advanced anal squamous cell carcinoma: results from the non-randomised, multicohort, multicentre, phase 2 KEYNOTE-158 study. Lancet Gastroenterol Hepatol. 2022 May;7(5):446-454. doi: 10.1016/S2468-1253(21)00382-4. Epub 2022 Feb 1. PMID 35114169
- [Derived] O'Malley DM, Bariani GM, Cassier PA, Marabelle A, Hansen AR, De Jesus Acosta A, Miller WH Jr, Safra T, Italiano A, Mileshkin L, Xu L, Jin F, Norwood K, Maio M. Pembrolizumab in Patients With Microsatellite Instability-High Advanced Endometrial Cancer: Results From the KEYNOTE-158 Study. J Clin Oncol. 2022 Mar 1;40(7):752-761. doi: 10.1200/JCO.21.01874. Epub 2022 Jan 6. PMID 34990208
- [Derived] Yap TA, Nakagawa K, Fujimoto N, Kuribayashi K, Guren TK, Calabro L, Shapira-Frommer R, Gao B, Kao S, Matos I, Planchard D, Chatterjee A, Jin F, Norwood K, Kindler HL. Efficacy and safety of pembrolizumab in patients with advanced mesothelioma in the open-label, single-arm, phase 2 KEYNOTE-158 study. Lancet Respir Med. 2021 Jun;9(6):613-621. doi: 10.1016/S2213-2600(20)30515-4. Epub 2021 Apr 6. PMID 33836153
- [Derived] Marabelle A, Fakih M, Lopez J, Shah M, Shapira-Frommer R, Nakagawa K, Chung HC, Kindler HL, Lopez-Martin JA, Miller WH Jr, Italiano A, Kao S, Piha-Paul SA, Delord JP, McWilliams RR, Fabrizio DA, Aurora-Garg D, Xu L, Jin F, Norwood K, Bang YJ. Association of tumour mutational burden with outcomes in patients with advanced solid tumours treated with pembrolizumab: prospective biomarker analysis of the multicohort, open-label, phase 2 KEYNOTE-158 study. Lancet Oncol. 2020 Oct;21(10):1353-1365. doi: 10.1016/S1470-2045(20)30445-9. Epub 2020 Sep 10. PMID 32919526
- [Derived] Piha-Paul SA, Oh DY, Ueno M, Malka D, Chung HC, Nagrial A, Kelley RK, Ros W, Italiano A, Nakagawa K, Rugo HS, de Braud F, Varga AI, Hansen A, Wang H, Krishnan S, Norwood KG, Doi T. Efficacy and safety of pembrolizumab for the treatment of advanced biliary cancer: Results from the KEYNOTE-158 and KEYNOTE-028 studies. Int J Cancer. 2020 Oct 15;147(8):2190-2198. doi: 10.1002/ijc.33013. Epub 2020 May 2. PMID 32359091
- [Derived] Strosberg J, Mizuno N, Doi T, Grande E, Delord JP, Shapira-Frommer R, Bergsland E, Shah M, Fakih M, Takahashi S, Piha-Paul SA, O'Neil B, Thomas S, Lolkema MP, Chen M, Ibrahim N, Norwood K, Hadoux J. Efficacy and Safety of Pembrolizumab in Previously Treated Advanced Neuroendocrine Tumors: Results From the Phase II KEYNOTE-158 Study. Clin Cancer Res. 2020 May 1;26(9):2124-2130. doi: 10.1158/1078-0432.CCR-19-3014. Epub 2020 Jan 24. PMID 31980466
- [Derived] Chung HC, Ros W, Delord JP, Perets R, Italiano A, Shapira-Frommer R, Manzuk L, Piha-Paul SA, Xu L, Zeigenfuss S, Pruitt SK, Leary A. Efficacy and Safety of Pembrolizumab in Previously Treated Advanced Cervical Cancer: Results From the Phase II KEYNOTE-158 Study. J Clin Oncol. 2019 Jun 10;37(17):1470-1478. doi: 10.1200/JCO.18.01265. Epub 2019 Apr 3. PMID 30943124
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26183&tenant=MT_MSD_9011